CLINICAL TRIAL: NCT04037371
Title: Effects of Environmental Temperature on Human White Adipose Tissue Thermogenic Capacity
Brief Title: Environmental Temperature and Human White Adipose Tissue
Status: Completed | Type: Observational
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Other Study IDs: 1. PET/CT & Tenv
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Obesity, Abdominal; Obese
Keywords: Cold exposure; white fat cells; thermoregulation; winter
MeSH Terms: conditions — Obesity; Obesity, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cold exposure — Participants were tested for white fat thermogenic activity against their environmental temperature exposure

SUMMARY:
Obesity is characterized by excessive white adipose tissue (WAT) that increases risk for disease. About 700 million adults are obese worldwide, designating the need of reducing excessive WAT in humans and subsequently the risk for disease. For this reason, previous research focused on the thermogenic capacity of white adipocytes in response to cold exposure. The investigators aimed to identify whether human WAT thermogenic activation could alter energy homeostasis and subsequently total body weight. The human WAT thermogenic capacity was assessed via Positron Emission Tomography/Computed Tomography (PET/CT) examination.

DETAILED DESCRIPTION:
PET/CT cooling protocol Participants recruited through an advertisement in local newspapers or by word of mouth. An initial appointment was made to inform participants about the study and determine eligibility. A health pre-screening was done by interview through a suitable medical history questionnaire. The investigators obtained written consent from 20 healthy (no chronic disease and/or being under medication treatment) and non-smoking adult men [age: 36.30±5.33 (years); Body Mass Index: 28.46±5.49 (kg/m2)].

On the day of the measurements the participants advised to transport themselves by car to the PET/CT Laboratory at 07:30 am, following at least a 12-hour fasting. At 8 am the participants consumed a meal consisted of 50% carbohydrates, 20% proteins and 30% fat to avoid a thermic effect of food on white adipose tissue (WAT) activity. Also, to avoid a thermic effect of food on the Resting Energy Expenditure (REE) measurement, the caloric value of the meal was 15% of the total energy requirements of each participant. The total energy requirements was calculated following previous methodology. At 14:00 pm participants underwent measurements for body height using a Seca (Hamburg, Germany) stadiometer, body weight using a precision scale (KERN & Sohn GmbH, Version 5.3, Germany) and Waist Hip Ratio using a tape measure. The investigators also measured blood pressure using a Standard Aneroid sphygmomanometer (Medisave, UK) according to standard guidelines. Blood glucose levels were determined via a Contour NEXT/ASCENSIA monitor. Participants who displayed blood glucose >140 mg/dl and blood pressure >140 mm/Hg were excluded from the study.

Immediately after the aforementioned measurements participants wore specific clothes (long-sleeve sweatshirt and sweatpants) that offered 0.49 clo insulation. Participants then undertook a REE assessment. Following the REE measurement participants remained in a sitting position in a cold room at 16-17ºC (humidity ~30-40%) for two hours. The room temperature and humidity were continuously monitored, while an investigator checked every 15 minutes participants muscle shivering status, according to previous methodology. The muscle shivering was tested using a scale, none (no tension of muscles reported), mild (slight muscle tonus in masseter muscle), moderate (real shivering in proximal muscles), severe (uncontrolled shivering in whole body). In case of moderate or severe shivering, participants were covered with a blanket for the next 15 minutes. After the first hour of cold exposure an appropriate dose - according to participants body weight - of F18 fludeoxyglucose (18F-FDG) was injected to the participants.

Following the 2-hour cooling protocol participants undertook the PET/CT examination. A Siemens Biograph 6 high resolution Erlangen Germany (2006) PET/CT was used to obtain images from the top of the skull to the upper third of the thigh. Six to eight bed positions (five minutes per bed position) were required.

White adipose tissue activity analysis WAT activity analysis (dorsolumbar region near vertebrae L3 and abdominal region) was performed by two independent trained physicians.

REE assessments for PET/CT cooling protocol REE assessments were conducted between 14:00 to 15:00 pm to comply with guidelines regarding the thermic effect of food on REE. The investigators have also instructed the participants to refrain from exercise, alcohol, and passive smoking in 72-hour prior to the measurements. REE was measured using an automated portable gas analyser (Oxycon Mobile, CareFusion, San Diego, USA) and the procedure was identical to the REE assessment for our UCP1 studies described above.

Environmental temperature (Tenv) recording Environmental data (ambient temperature) were obtained from Weather Underground (www.wunderground.com). Tenv was recording between January 2017 and March 2019. For the latter periods, the investigators obtained daily mean air temperature from the closest weather station operated near the area participants lived; the weather station Eleftherios Venizelos international station, Athens, Greece (37.93 °N, 23.93 °E) at an elevation of 94m.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult men
* no chronic disease
* not being under medication treatment
* non-smoking individuals
* non-regular exercisers individuals

Exclusion Criteria:

* non-adult men
* women
* chronic disease
* being under medication treatment
* smokers
* regular exercisers

Max Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 20 healthy adult men [age: 36.30±5.33 (years); Body Mass Index: 28.46±5.49 (kg/m2)]
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Correlation between white adipose tissue activity and environmental temperature. Mean differences in white adipose tissue activity between those participants who were assessed in winter and those who were assessed in summer. | An overall of 10 hours of an assessment period that including two hours of cold exposure, 30 minutes of resting energy expenditure and 40 minutes of PET/CT assessments
  White adipose tissue activity was assessed using a PET/CT examination to calculate the standardized uptake value (SUV) in dorsolumbar region near vertebrae L3 and abdominal region. Daily environmental temperature was obtained in degrees Celsius from the Weather Underground (www.wunderground.com) webpage for the period between January 2017 and February 2019

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Flouris, PhD, Principal Investigator — FAME Laboratory, Department of Exercise Science, University of Thessaly
Locations (1):
- Petros Dinas, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided